CLINICAL TRIAL: NCT03649269
Title: Eryngium Heterophyllum + Amphipterygium Adstringens Tea Effect on Triglyceride Levels
Brief Title: PC-300 Tea Effect on Triglyceride Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciprés Grupo Médico CGM SC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/02
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Hypertriglyceridemia
Keywords: Eryngium heterophyllum; Amphipterygium adstringens; tea
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Teas, Herbal; Bezafibrate

STUDY DESIGN:
Intervention Model Description: Voluntary subjects were assigned sequentially into two treatment groups: 1) fibrate (bezafibrate) 200 mg/day, and 2) PC-300 tea, one cup half an hour before eating.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PC-300 tea (Experimental): Patients that received the Eryngium heterophyllum + Amphipterygium adstringens tea, one cup half an hour before eating.
  Interventions: Dietary Supplement: PC-300 tea.
- Bezafibrate (Active Comparator): Patients that received fibrate (bezafibrate) 200 mg/day.
  Interventions: Drug: Bezafibrate

INTERVENTIONS:
Dietary Supplement: PC-300 tea. — Patients had to drink one cup of the tea half an hour before breakfast, main meal and dinner.
  Other Names: Herbal tea
  Arms: PC-300 tea
Drug: Bezafibrate — Patients were prescribed 200 mg/day at night.
  Other Names: Bezalip
  Arms: Bezafibrate

SUMMARY:
Herbal medicine represents an alternative for treating dyslipidemia. The aim of this project was to evaluate the PC-300 tea (Eryngium heterophyllum egelm + Amphipterygium adstringens) against hypertriglyceridemia.

Baseline samples of serum total cholesterol and triglycerides were obtained and measured again after 1 month of treatment with the following two alternatives: 1) PC-300, one cup half an hour before eating, and 2) bezafibrate 200 mg/d.

DETAILED DESCRIPTION:
It was a descriptive, prospective, longitudinal, and comparative clinical study developed at Ciprés Grupo Médico S.C. (CGM), Toluca, Mexico, from January 2014 to December 2014.

Patients with hypertriglyceridemia were invited to participate in the study. Voluntary subjects were assigned sequentially into two treatment groups: 1) fibrate (bezafibrate) 200 mg/day, and 2) PC-300 tea, one cup half an hour before eating.

Patients were measured (m) and weighed (kg) (Obi, México). Body mass index (BMI) was calculated as weight (kg) divided by height (m) squared. Blood pressure was measured with a calibrated sphygmomanometer (Welch Allyn, USA) after 5 min of rest.

All of the patients were given a low lipid diet. Calculated kcal were based on ideal weight minus 200 kcal/day if overweight.

Results were expressed as mean ± Standard deviation (SD). Differences between initial vs. final values were compared with the Mann-Whitney U test. The normality hypothesis was tested using the Kolmogorov-Smirnov test. A p value of <0.05 was considered significant. All tests were performed with the SPSS ver. 23 statistical software program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertriglyceridemia, aged >18 years and with an educational level at least of primary school.

Exclusion Criteria:

* Patients with hepatic disease and those missing an appointment during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Triglycerides serum levels. | One month.
  The triglycerides serum levels were measured at the recruiting moment and after one month..

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Mendieta Zerón, PhD., Principal Investigator — Ciprés Grupo Médico

IPD SHARING:
Plan to Share IPD: Undecided
With this first study researcher are not planning to share the IPD.